CLINICAL TRIAL: NCT03905135
Title: A Phase 1 Study of Interleukin-15 in Combination With Avelumab (Bavencio) in Relapsed/Refractory Mature T-cell Malignancies
Brief Title: Interleukin-15 (IL-5) in Combination With Avelumab (Bavencio) in Relapsed/Refractory Mature T-cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Conlon, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190076; 19-C-0076
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Results first posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Peripheral T-cell Lymphoma NOS; Mycosis Fungoides; Sezary Syndrome; Anaplastic Large Cell Lymphoma
Keywords: T-cell Lymphoproliferative Disorder; Cutaneous T-Cell Lymphoma; Anti-PD-L1 monoclonal antibody; Antibody Dependent Cellular Cytotoxicity (ADCC)
MeSH Terms: conditions — Lymphoma, T-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell, Cutaneous | interventions — Interleukin-15; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1- Experimental Treatment: Dose Escalation (Experimental): Interleukin-15 (IL-15) by continuous intravenous (civ) infusion at escalating doses of 1, 2, 3 and 4 mcg/kg/day on days 1-5 of each 28-day cycle (max 6 cycles) with avelumab by intravenous (IV) infusion at a dose of 10mg/kg on Day 8 and 22 of each cycle, to determine maximum tolerated dose (MTD)
  Interventions: Drug: rhIL-15; Biological: Avelumab
- 2- Experimental Treatment: Dose Expansion (Experimental): Interleukin-15 (IL-15) by continuous intravenous (civ) infusion at the maximum tolerated dose (MTD) on days 1-5 of cycles 1-6 with avelumab at 10mg/kg on Day 8 and 22 of each cycle
  Interventions: Drug: rhIL-15; Biological: Avelumab

INTERVENTIONS:
Drug: rhIL-15 — Interleukin-15 (IL-15) will be administered by continuous intravenous infusion in a dose-escalation fashion with a starting dose level of 1 mcg/kg/day, a second dose level of 2 mcg/kg/day, a third dose level at 3 mcg/kg/day, and a fourth dose level at 4 mcg/kg/day on days 1-5 of each of six cycles.
  Other Names: Recombinant human Interleukin-15
  Arms: 1- Experimental Treatment: Dose Escalation
Drug: rhIL-15 — Interleukin-15 (IL-15) will be administered by continuous intravenous infusion at the maximum tolerated dose (MTD) or maximum administered dose (MAD) on days 1-5 of each of six cycles
  Other Names: Recombinant human Interleukin-15
  Arms: 2- Experimental Treatment: Dose Expansion
Biological: Avelumab — Avelumab (intravenous (IV) over 1 hour) will be administered at a dose of 10 mg/kg on days 8 and 22 of each of six cycles.
  Other Names: Bavencio

SUMMARY:
Background:

Some T-cell lymphomas and leukemias do not respond to standard treatment. Researchers hope to develop a treatment that works better than current treatments.

Objective:

To test if interleukin (IL-5) combined with avelumab is safe and effective for treating certain cancers.

Eligibility:

People ages 18 and older with relapsed T-cell leukemias and lymphomas for which no standard treatment exists or standard treatment has failed

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood, urine, heart, and lung tests
* Possible tumor biopsy
* Bone marrow biopsy: A small needle will be inserted into the hipbone to take out a small amount of marrow.
* Computed tomography (CT) or positron emission tomography (PET) scans and magnetic resonance imaging (MRI): Participants will lie in a machine that takes pictures of the body.

Participants will get the study drugs for 6 cycles of 28 days each. They will have a midline catheter inserted: A tube will be inserted into a vein in the upper chest. They will get Interleukin-15 (IL-5) as a constant infusion over the first 5 days of every cycle. They will get avelumab on days 8 and 22 of each cycle. They will be hospitalized for the first week of the first cycle.

Participants will have tests throughout the study:

* Blood and urine tests
* Another tumor biopsy if their disease gets worse
* Scans every 8 weeks
* Possible repeat MRI
* Another bone marrow biopsy at the end of treatment, if there was lymphoma in the bone marrow before treatment, and they responded to treatment everywhere else.

After they finish treatment, participants will have visits every 60 days for the first 6 months. Then visits will be every 90 days for 2 years, and then every 6 months for 2 years. Visits will include blood tests and may include scans.

DETAILED DESCRIPTION:
Background:

Mature T-cell cancers are a phenotypically heterogeneous group of malignancies which constitute 10-15% of all non-Hodgkin lymphomas (NHL). Patients with relapsed/refractory T cell lymphomas have limited therapeutic options, making new therapeutic approaches extremely important.

The immunologic effects of recombinant human Interleukin-15 (rhIL-15), a stimulatory cytokine that promotes the differentiation and activation of NK cells, monocytes and long-term cluster of differentiation 8 (CD8) + memory T-cells, has been assessed in several Phase 1 trials in cancer patients.

Avelumab is an anti-programmed death ligand-1 (PD-L1) fully human immunoglobulin G1 (IgG1) antibody that inhibits programmed cell death protein 1 (PD1)/PD-L1 interactions while leaving the PD1/programmed cell death ligand 2 (PD-L2) pathway intact and enhances immune activation against tumor cells. It has received United States (U.S.) Food and Drug Administration (FDA) accelerated approval for the treatment of patients with metastatic Merkel cell carcinoma (MCC) and urothelial carcinoma.

Unlike other approved anti-PD-L1/PD1 antibodies, avelumab induces lysis of tumor cells via antibody-dependent cell-mediated cytotoxicity (ADCC), indicating an additional mechanism of action. However, avelumab has not shown ADCC against normal immune cell subsets in humans.

A significant number of T-cell malignancies express PD-L1, and since the anti-PD-L1 antibody avelumab has shown ADCC activity in vitro, agents that may enhance ADCC by increasing number and activity of Fc-binding effector cells such as rhIL15 could improve efficacy of avelumab in these diseases.

Objectives:

To determine the safety and toxicity profile and the maximum tolerated dose (MTD) of continuous intravenous infusion (civ) recombinant human interleukin-15 (rhIL-15) administration in combination with standard intravenous (IV) avelumab treatment

Eligibility:

Age >= 18 years of age

Eastern Cooperative Oncology Group (ECOG) performance status of <= 1

Histologically or cytologically confirmed relapsed and/or refractory T-cell lymphoma other than adult T-cell leukemia/lymphoma (ATLL), angioimmunoblastic T-cell lymphoma (AITL), peripheral T-cell lymphoma T follicular helper phenotype (PTCL-TFH) and enteropathy-associated T-cell lymphoma (EATL).

Adequate organ and marrow function

Design:

Open-label, single-center, non-randomized Phase 1 study

Standard 3 + 3 design will be used to determine the MTD of dose-escalated rhIL-15 with fixed dose avelumab with a small expansion cohort at the MTD

Maximum 6 cycles (28-day cycle) of combination therapy

To explore all dose levels, including further evaluation in a dose expansion cohort, the accrual ceiling will be set at 30 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically proven relapsed/refractory T-cell lymphoma other than adult T-cell leukemia/lymphoma (ATLL), angioimmunoblastic T-cell lymphoma (AITL), peripheral T-cell lymphoma T follicular helper phenotype (PTCL-TFH), or enteropathy-associated T-cell lymphoma (EATL), confirmed by the Laboratory of Pathology, National Cancer Institute (NCI)
* Patients with CD30 (also known as TNFRSF8) + mycosis fungoides/Sezary syndrome (MF/SS) or CD30+ anaplastic large cell lymphoma (ALCL) must have relapsed after or become intolerant to treatment with brentuximab vedotin.
* A formalin fixed tissue block or 15 slides of tumor sample (archival or fresh) must be available for performance of correlative studies. NOTE: Patients must be willing to have a tumor biopsy if prior tissue or adequate archival tissue is not available (i.e., post-enrollment and prior to treatment).
* Disease must be measurable with at least one measurable lesion by response evaluation criteria in lymphoma (RECIL) 2017 or Modified Severity-Weighted Assessment Tool (mSWAT) criteria or have an abnormal clonal T-cell population detectable by peripheral blood flow cytometry
* Age greater than or equal to 18 years

NOTE: Because no dosing or adverse event data are currently available on the use of rhIL-15 in combination with avelumab in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials

* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1
* Adequate organ and marrow function as defined:

  * Absolute neutrophil count greater than 1,000/mcL
  * Absolute lymphocyte count greater than or equal to 500/mcL
  * Hemoglobin greater than or equal to 9 g/dL
  * Platelets greater than 100,000/mcL
  * Total bilirubin less than or equal to 1.5 X institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) Serum glutamic oxaloacetic transaminase (SGOT)/Alanine aminotransferase (ALT) Serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 X institutional ULN
  * Serum creatinine less than or equal to 1.5 X institutional ULN OR
  * Creatinine clearance greater than or equal to 50 mL/min/1.73 m^2 for patients with creatinine levels greater than 1.5 institutional ULN
* Negative serum or urine pregnancy test at screening for women of childbearing potential (WOCBP)

NOTE: WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal. WOCBP must have a negative pregnancy test (human chorionic gonadotropin (HCG) blood or urine) during screening.

* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 30 days after completion of rhIL-15 and avelumab administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Patients with the following T-cell leukemias/lymphomas: adult T-cell leukemia/lymphoma (ATLL), angioimmunoblastic T-cell lymphoma (AITL), peripheral T-cell lymphoma T follicular helper phenotype (PTCL-TFH), and enteropathy-associated T-cell lymphoma (EATL).
* Chemotherapy and anti-tumor antibodies within 4 weeks (6 weeks for nitrosoureas or mitomycin C); other tumor-directed systemic therapy and radiation therapy within 2 weeks.
* Persisting toxicity related to prior therapy of grade > 1, with the exception of the following: alopecia, sensory neuropathy grade less than or equal to 2, or other grade less than or equal to 2 not constituting a safety risk based on investigator's judgment
* Patients who are receiving any other investigational agents
* Patients who have had prior therapy with any antibody/drug targeting programmed cell death protein 1 (PD-1)/programmed death-ligand 1 (PD-L1) Tcell coregulatory proteins (immune checkpoints)
* Current use of immunosuppressive medication, EXCEPT for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses less than or equal to 10 mg/day of prednisone or equivalent; or,
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography (CT) scan premedication)
* Patients with known central nervous system (CNS) involvement should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients with previous malignant disease other than the target malignancy within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ
* Patients with history of any organ transplantation, including allogenic stem cell transplantation
* Received a live vaccine within 4 weeks of the first dose of avelumab. Vaccination with a live vaccine while on trial is prohibited. NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Patients with history of allergic reactions attributed to compounds of similar chemical or biologic composition to recombinant human Interleukin-15 (rhIL-15) or avelumab
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring systemic therapy, or psychiatric illness/social situations that would limit compliance with study requirements
* Inability or refusal to practice effective contraception during therapy or the presence of pregnancy or active breastfeeding. Based on its mechanism of action, avelumab can cause fetal harm when administered to a pregnant woman. Animal studies have demonstrated that inhibition of the PD-1/PD-L1 pathway can lead to increased risk of immune-mediated rejection of the developing fetus resulting in fetal death. These potential risks may also apply to other agents used in this study
* Patients with active bacterial infections, documented human immunodeficiency virus (HIV) infection or positive screening serology, polymerase chain reaction (PCR) evidence for active or chronic hepatitis B or hepatitis C, or positive screening hepatitis B virus (HBV)/hepatitis C virus (HCV) serology without documentation of successful curative treatment
* Patients with active or history of any autoimmune disease, unrelated to their malignancy, including asthma requiring chronic inhaled or oral corticosteroids, or with history of asthma requiring mechanical ventilation; patients with a history of mild asthma that are on or can be switched to non-corticosteroid bronchodilator regimens are eligible
* Cardiovascular disease: Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (greater than or equal to New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Conlon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
  In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely. Genomic data will be available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).
  Genomic data will be made available via database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Dubois SP, Miljkovic MD, Fleisher TA, Pittaluga S, Hsu-Albert J, Bryant BR, Petrus MN, Perera LP, Muller JR, Shih JH, Waldmann TA, Conlon KC. Short-course IL-15 given as a continuous infusion led to a massive expansion of effective NK cells: implications for combination therapy with antitumor antibodies. J Immunother Cancer. 2021 Apr;9(4):e002193. doi: 10.1136/jitc-2020-002193. PMID 33883258
- [Derived] Waldmann TA, Dubois S, Miljkovic MD, Conlon KC. IL-15 in the Combination Immunotherapy of Cancer. Front Immunol. 2020 May 19;11:868. doi: 10.3389/fimmu.2020.00868. eCollection 2020. PMID 32508818
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0076.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled on dose level 3, dose level 4, and expansion cohort because the manufacturer withdrew support due to low enrollment.
Groups:
- Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab: Interleukin-15 (IL-15) will be administered by continuous intravenous infusion in a dose-escalation fashion with a starting dose level of 1 mcg/kg/day on days 1-5 of each of six cycles.
  Avelumab (intravenous (IV) over 1 hour) will be administered at a dose of 10 mg/kg on days 8 and 22 of each of six cycles.
- Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab: Interleukin-15 (IL-15) will be administered by continuous intravenous infusion in a dose-escalation fashion with a second dose level of 2 mcg/kg/day on days 1-5 of each of six cycles.
  Avelumab (intravenous (IV) over 1 hour) will be administered at a dose of 10 mg/kg on days 8 and 22 of each of six cycles.
Period: Dose Escalation
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
Started | 6 | 2
Completed | 1 | 0
Not Completed | 5 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Progressive disease | 3 | 1
Not completed — Intercurrent illness | 1 | 0
Period: Dose Expansion
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (5.26) | 57.9 (12.45) | 59.33 (6.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Interleukin 15
Description: The MTD is the dose level at which no more than 1 of up to 6 participants experience a dose-limiting toxicity (DLT) during the DLT evaluation window(s), or the dose below that at which at least 2 (of ≤6) participants have DLT. A dose-limiting toxicity (DLT) is defined as: any grade 3, 4, or 5 toxicity, if not incontrovertibly due to disease progression or an extraneous cause, and deemed possibly, probably or definitely related to interleukin-15 (IL-5) by the principal investigator (PI) or designee during the first 28 days of treatment. Grade 3 is severe. Grade 4 is life threatening. Grade 5 is death related to adverse event.
Time Frame: First 28 days of treatment
Measure: Number; unit: mcg/kg
Groups:
- Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab: Interleukin-15 (IL-15) will be administered by continuous intravenous infusion in a dose-escalation fashion with a starting dose level of 1 mcg/kg/day on days 1-5 of each of six cycles.
- Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab: Interleukin-15 (IL-15) will be administered by continuous intravenous infusion in a dose-escalation fashion with a second dose level of 2 mcg/kg/day on days 1-5 of each of six cycles.
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
Number analyzed (Participants) | 6 | 2
mcg/kg | NA — The MTD was not found because the study was halted due to manufacturer withdrawal of support for low enrollment. | NA — The MTD was not found because the study was halted due to manufacturer withdrawal of support for low enrollment.

2. Secondary Outcome: Mean Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, or death, whichever occurs first. Disease relapse is Disease progression is >20% increase in the sum of longest diameters of target lesions or appearance of a new lesion assessed by the Response Evaluation Criteria in Lymphoma (RECIL) 2017 criteria.
Time Frame: From study opening through May 2022 when the study was completed with a maximum follow up of approximately 2 years and 11 months for any participant.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
Number analyzed (Participants) | 6 | 2
Days | 303 (242) | 61.5 (55.9)

3. Secondary Outcome: Mean Event-free Survival (EFS)
Description: EFS is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, alternative therapy for lymphoma given (such as radiation), or death, whichever occurs first, and was estimated using Kaplan-Meier curves along with a 95% confidence interval. Disease relapse is Disease progression is >20% increase in the sum of longest diameters of target lesions or appearance of a new lesion assessed by the Response Evaluation Criteria in Lymphoma (RECIL) 2017 criteria.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
Number analyzed (Participants) | 6 | 2
Days | 176 (140) | 33.54 (0.98)

4. Secondary Outcome: Mean Overall Survival (OS)
Description: OS is defined as the time from the date of study enrollment until time of death from any cause and was estimated using Kaplan-Meier curves along with a 95% confidence interval.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
Number analyzed (Participants) | 6 | 2
Days | 529 (345) | 300 (430)

5. Secondary Outcome: Overall Response in Participants With Greater Than or Equal to 50% Programmed Death-ligand 1 (PD-L1) Expressing Tumor Cells
Description: Response was assessed by the Response Evaluation Criteria in Lymphoma (RECIL) 2017 criteria and reported along with a 95% confidence interval. Complete response is complete disappearance of all target lesions. Partial response is ≥30% decrease in the sum of longest diameters of target lesions but not a complete response. Minor response is ≥10% decrease in the sum of longest diameters of target lesions but not a partial response. Stable disease is <10% decrease or ≤20% increase in the sum of longest diameters of target lesions. Disease progression is >20% increase in the sum of longest diameters of target lesions or appearance of a new lesion.
Time Frame: From the time the subject began protocol treatment until end of treatment, progression or start of another therapy or approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
Number analyzed (Participants) | 6 | 2
Participants
  Partial Response | 2 | 0
  Progressive Disease | 2 | 2
  Stable Disease | 2 | 0
  Minor Response | 0 | 0

6. Secondary Outcome: Number of Participants With Overall Best Response
Description: OR is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Complete response is complete disappearance of all target lesions. Partial response is ≥30% decrease in the sum of longest diameters of target lesions but not a complete response. Minor response is ≥10% decrease in the sum of longest diameters of target lesions but not a partial response. Stable disease is <10% decrease or ≤20% increase in the sum of longest diameters of target lesions. Disease progression is >20% increase in the sum of longest diameters of target lesions or appearance of a new lesion assessed by the Response Evaluation Criteria in Lymphoma (RECIL) 2017 criteria.
Time Frame: 6 cycles (each cycle is 28 days) - approximately 168 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
Number analyzed (Participants) | 6 | 2
Participants
  Complete Response | 0 | 0
  Partial Response | 2 | 0
  Minor Response | 0 | 0
  Stable Disease | 2 | 0
  Progressive Disease | 2 | 2

7. Secondary Outcome: Mean Duration of Response (DOR)
Description: DOR is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is recorded first) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started), death, or, in the absence of progressive disease (PD), date of last assessment. The response rate was assessed by the Response Evaluation Criteria in Lymphoma (RECIL) 2017 criteria and reported along with a 95% confidence interval. Complete response is complete disappearance of all target lesions. Partial response is ≥30% decrease in the sum of longest diameters of target lesions but not a complete response. Disease progression is >20% increase in the sum of longest diameters of target lesions or appearance of a new lesion.
Time Frame: From the time that response to therapy is first documented until progressive disease is observed or the subject is lost to follow-up or approximately 2 years.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
Number analyzed (Participants) | 6 | 2
Days | 107 (115) | NA (NA) — Cannot report because none in dose level 2 had a partial response or complete response.

8. Other Pre Specified Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: A dose-limiting toxicity (DLT) is defined as: any grade 3, 4, or 5 toxicity if not incontrovertibly due to disease progression or an extraneous cause, and deemed possibly, probably or definitely related to interleukin-15 (IL-5) or avelumab by the principal investigator (PI) or designee during the first 28 days of treatment. Grade 3 is severe. Grade 4 is life threatening. Grade 5 is death related to adverse event.
Time Frame: First 28 days of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
Number analyzed (Participants) | 6 | 2
Participants | 1 | 1

9. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 21 months and 18 days for the dose level 1 and 3 months and 19 days for the dose level 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
Number analyzed (Participants) | 6 | 2
Participants | 6 | 2

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 21 months and 18 days for the dose level 1 and 3 months and 19 days for the dose level 2.
Description: Three participants died from disease progression during the long-term survival follow-up phase of the study (they were only being called once every 3 months to check to see if they died and to learn of new cancer treatments). We were no longer tracking adverse events (AEs) at the time of death, thus only one death from progressive disease is listed in the serious adverse events table below.
Groups:
- Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab; Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab: Interleukin-15 (IL-15) will be administered by continuous intravenous infusion in a dose-escalation fashion with a starting dose level of 1 mcg/kg/day, a second dose level of 2 mcg/kg/day, a third dose level at 3 mcg/kg/day, and a fourth dose level at 4 mcg/kg/day on days 1-5 of each of six cycles.
  Avelumab (intravenous (IV) over 1 hour) will be administered at a dose of 10 mg/kg on days 8 and 22 of each of six cycles.
Arm/Group | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab
All-Cause Mortality (participants affected / at risk) | 3/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 6/6 | 0/2
Other Adverse Events (participants affected / at risk) | 3/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab (N=6) | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab (N=2)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation - Dose Level 1, 1mcg/kg Interleukin-15 With 10 mg Avelumab (N=6) | Dose Level 2, 2mcg/kg Interleukin-15 With 10 mg Avelumab (N=2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (6) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, neutrophilia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (3) | 0 (0)
Chills (General disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 2 (4) | 1 (3)
Generalized edema (General disorders) | 1 (2) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (5) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (6) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT03905135/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT03905135/ICF_001.pdf